CLINICAL TRIAL: NCT05044169
Title: Efficacy and Safety of Broncho-Vaxom in Reducing Recurrence in Children With Steroid-sensitive Nephrotic Syndrome: Prospective, Randomized Controlled, Multicenter Clinical Study
Brief Title: Efficacy and Safety of Broncho-Vaxom in the First Episode of Pediatric Idiopathic Nephrotic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fang Deng (Other)
Responsible Party: Sponsor-Investigator, Fang Deng, PI, Anhui Provincial Children's Hospital
Organization: Anhui Provincial Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnhuiPCH
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Nephrotic Syndrome in Children
Keywords: relapse; infection
MeSH Terms: conditions — Recurrence; Infections | interventions — Broncho-Vaxom

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Broncho-Vaxom (Experimental): Intervention
  Interventions: Drug: Broncho-Vaxom

INTERVENTIONS:
Drug: Broncho-Vaxom — administration for 6 months after remmission
  Other Names: OM-85BV

SUMMARY:
The main objective is to demonstrate, from the initial episode of nephrotic syndrome (NS) in children with standard prednisolone treatment, once complete remission has occurred, that the use of Broncho-Vaxom (administration for 6 months) may reduce the risk of subsequent relapse during 12-month of follow-up.

DETAILED DESCRIPTION:
NS is the most frequent glomerular disease in children. Between 80% and 90% of children with steroid-sensitive nephrotic syndrome (SSNS) will relapse following an initial response to corticosteroids. Half of these children will experience frequent relapses (FRNS) or become steroid-dependent (SDNS).

Infection is the most common and serious complication in children with NS. More than 80% patients had infections before relapse. The results of multiple observational studies and randomized control trials have shown that Broncho-Vaxom, a lysate of 8 common bacterial respiratory pathogens, is safe and effective to prevent infections in children. To the investigators' knowledge, Broncho-Vaxom has never been investigated for the initial episode of NS with the aim to reduce the subsequent risk of relapse that is a major concern in the management of children with NS.

Children aged 1-18 years with the first episode of the SSNS will be treated with Broncho-Vaxom for 6 months. The prednisolone at a dose of 2 mg/kg per day (maximum 60 mg in single or divided doses) for 6 weeks, followed by 1.5 mg/kg (maximum 40 mg) as a single morning dose on alternate days for the next 6 weeks; therapy is then discontinued.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children between 1 and 18 years with Steroid-Sensitive Nephrotic Syndrome. 2. Estimated glomerular filtration rate (eGFR) ≥90 ml/min per 1.73 m2 at study entry.

  3. Remission at study entry. 4.No immunosuppressive agents have been used within 3 months of enrollment, except for the use of corticosteroid to treat nephrotic syndrome.

  5. Provision of consent by a legal representative (parents or legal guardians) using a document approved by the institutional review board after receiving an adequate explanation regarding the implementation of this clinical trial. For children/youth ages 10-18, written assent is required using age-appropriate and background-appropriate documents.

Exclusion Criteria:

* 1.Diagnosis of secondary NS 2.Patients showing one of the following abnormal clinical laboratory values: leukopenia (white blood cell count ≤3.0*109/L); moderate and severe anemia (hemoglobin <9.0g/dL); thrombocytopenia (platelet count <100*1012/ L); positivity of autoimmunity tests (ANA, Anti DNA antibody, ANCA) or reduced C3 levels; Positive for hepatitis B surface (HBs) antigen, HBs antibody, hepatitis B core (HBc) antibody, or hepatitis C virus (HCV) antibody ; Positive for HIV antibody; Alanine aminotransferase (ALT) > 2.5× upper limit of normal value. Aspartate aminotransferase (AST) > 2.5× upper limit of normal value.

  3. Presence or history of severe or opportunistic infections within 6 months before assignment; Presence of active tuberculosis or with a history of tuberculosis or in whom tuberculosis is suspected; Presence or history of chronic active infections such as Epstein-Barr virus and CMV virus; presence or history of active hepatitis B or hepatitis C or hepatitis B virus carrier. Presence of human immunodeficiency virus (HIV) infection or other active viral infections.

  4. History of angina pectoris, cardiac failure, myocardial infarction, or serious arrhythmia，or poorly controlled hypertension 5. Presence or history of autoimmune diseases or vascular purpura. 6. Presence or history of malignant tumor 7. History of organ transplantation (excluding corneal and hair transplants). 8. Patients with a known allergy to steroid and their excipients or to Broncho-Vaxom 9. Assessed to be unfit for participation by the investigators

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
1-year relapse-free survival rate | 1-year period after randomization
  The rate of no relapse within 1 year

SECONDARY OUTCOMES:
Time to relapse (days) | 1-year period after administration of Broncho-Vaxom therapy
  Number of days from randomization to occurrence of first relapse
Proportion of patients with a relapse | 6 months period after administration of Broncho-Vaxom therapy
  The proportion of patients with relapse
The effect of Broncho-Vaxom on peripheral blood B cell subsets and T cell subsets to highlight biomarkers useful for monitoring response to Broncho-Vaxom treatment. | 1-year period after administration of Broncho-Vaxom therapy
  Using fluorescence-activated cell sorting (FACS), peripheral blood B cell subsets and T cell subsets will be measured as at baseline, before and after infusion of Broncho-Vaxom at 3,6,9,12 months, and when relapse.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1-year period after administration of Broncho-Vaxom therapy
  It is a binary variable (1/0). The varibale would be setted as "1" if any adverse events occours including cough, diarrhea, abdominal pain, skin rashes, hives, swelling, eyelid/facial swelling, nausea, vomiting, systemic skin rashes, itching, fatigue, peripheral swelling, angioedema, etc. Adverse events will be graded according to the Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Deng, PhD.MD., Principal Investigator — Anhui Provincial Children's Hospital